CLINICAL TRIAL: NCT02197182
Title: An Open-Label, Randomized Study to Determine the Safety and Efficacy of LUXSOL(TM) Cream for the Treatment of Bacterial Vaginosis: A Proof of Concept Study
Brief Title: LUXSOL(TM) Topical Cream for the Treatment of Symptomatic Bacterial Vaginosis; A Proof of Concept Study
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Not for safety reasons
Sponsor: CDA Research Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDA 0801
Record Dates: First submitted 2014-07-20; First posted 2014-07-22 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-03

CONDITIONS: Bacterial Vaginosis (BV)
Keywords: Bacterial Vaginosis (BV); Amsel's criteria; Pap smear
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LUXSOL Cream (Experimental): LUXSOL Cream is a copper containing cream to be administered intravaginally before bedtime for 10 consecutive nights.
  Interventions: Drug: LUXSOL copper containing cream
- Metronidazole cream (Active Comparator): Metronidazole cream is the active comparator drug to be self-administered intravaginally each night before bedtime for 10 consecutive nights. Dosage is per package insert.
  Interventions: Drug: Metronidazole gel

INTERVENTIONS:
Drug: LUXSOL copper containing cream — Active comparator arm
  Other Names: LUXSOL Topical Cream
  Arms: LUXSOL Cream
Drug: Metronidazole gel — Active comparator for treatment of bacterial vaginosis
  Other Names: Metrogel
  Arms: Metronidazole cream

SUMMARY:
LUXSOL Cream may be useful for the treatment of bacterial Vaginosis. In this study, LUXSOL Cream is compared to a control arm group using metronidazole cream. LUXSOL is administered intravaginally for 10 days, each evening before bedtime to treat bacterial Vaginosis..

DETAILED DESCRIPTION:
LUXSOL Topical Cream is a copper containing topical cream indicated for the treatment of bacterial vaginosis (BV). The study is an open-label, randomized, controlled study comparing LUXSOL Cream to Metrogel in patients with a diagnosis of BV. The investigational product or the comparator product will be self-administered by the patient for 10 consecutive nights. A successful patient outcome is cured BV at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject agrees to participate and signs informed consent
* Female age 18 or older
* Subject has clinical BV with 4 of 4 Amsel's criteria
* Off-white (milky or gray), thin, adherent, homogenous discharge with minimal or absent pruritus and inflammation of the vulva and vagina
* Presence of 'clue cells' >/=20% of the total epithelial cells on microscopic examination of the saline 'wet mount.'
* Virginal secretion pH of >4.5
* A fishy odor of the vaginal discharge with the addition of a drop of 10% KOH (i.e. a positive 'whiff test')
* Subject agrees to refrain from use of douches, intravaginal products for treatment period
* Subject agrees to refrain from taking oral or intravaginal antibiotics or antifungal agents during entire study period
* Subject agrees to refrain from vaginal intercourse during treatment period.

Exclusion Criteria:

* Subject has another infectious or noninfectious cause of vulvovaginitis
* Subject has another vaginal or vulvar condition that would confound the determination of study endpoints.
* Subject has received antifungal or antimicrobial therapy (systemic or intravaginal) within the last 14 days prior to enrollment.
* Subject is under treatment for cervical intra-epithelial neoplasia or cervical carcinoma
* Subject is known to be HIV positive
* Subject has a positive pregnancy test
* Subject has any abnormal anatomy or pathology of the vagina
* Subject has untreated sexually transmitted disease
* Subject is currently having menstrual period or may have her period during treatment days.
* Subject's PAP smear >/= to LSIL
* Subjects with known sensitivity or allergic reactions to copper or Metronidazole vaginal gel
* Subject has known Wilson's disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Presence or absence of bacterial vaginosis at the end of the study | 30 days
  Patients will be assessed at day 30 for the presence or absence of bacterial Vaginosis (BV). Absence of BV will be considered a cure.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Harper University Hospital Department of Infectious Diseases, Detroit, Michigan
  - Temple University Hospital Department of OB/GYN, Philadelphia, Pennsylvania